CLINICAL TRIAL: NCT01441986
Title: A Phase IIa, Double-blind, Placebo-controlled, Randomised, Fourfold Crossover Study to Investigate the Glucose Lowering Effects of Dextromethorphan and Amantadine in Subjects With Type 2 Diabetes Mellitus (T2DM) After an Oral Glucose Tolerance Test
Brief Title: Dextromethorphan, Amantadine and Glucose Homeostasis in Diabetes Subjects
Acronym: DXM/AMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0533-DXM
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dextromethorphan; amantadine; blood glucose lowering effect; oral glucose tolerance test
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dextromethorphan; Amantadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dextromethorphan hydrobromide — Dextromethorphan hydrobromide•1 H2O; 30 mg; hard capsules; single, oral dose.
  Other Names: Dextromethorphan, Ratiopharm GmbH
Drug: Amantadine — Amantadine hydrochloride 100 mg; tablets; single, oral dose.
  Other Names: Amantadine, STADA Arzneimittel AG.
Drug: Pacebo 1 (placebo for Amantadine) — Talets for oral use; single dose.
  Other Names: P-Tabletten weiß 10 mm Lichtenstein, Winthrop Arzneimittel.
Drug: Placebo 2 (fo Dextromethorphan) — Capsles for oral administration; single dose.
  Other Names: Empty capsules, Capsugel Bornem Belgium.

SUMMARY:
The purpose of this trial is to demonstrate that dextromethorphan (DXM) and amantadine compared to placebo exert blood glucose (BG) lowering effects following an oral glucose tolerance test (OGTT) in male subjects with T2DM.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is characterized by hyperglycemia due to an impaired insulin activity (insulin resistance) or a reduced insulin production by the pancreas. The restoration of adequate insulin secretion represents one of the goals of several antidiabetic therapies such as sulfonylureas or incretin mimetics. Lowering blood glucose in type 2 diabetes mellitus (T2DM) prevents complications, microvascular complications in particular. Weight reduction is also a fundamental target in the treatment of T2DM; however, achieving weight loss through lifestyle measures is difficult, and the problem of obesity is often exacerbated by therapy with glucose-lowering agents such as insulin, that cause weight gain.

Pancreatic ß- cells are part of the pancreatic islets, of which 1-2 millions are located within the human pancreas. Interestingly, pancreas function is controlled in part by the central nervous system and ß- cells have many features in common with neurons, including the expression of tyrosine hydroxylase (TH), neural guidance molecules, such as Eph receptors and ephrins, neural cell adhesion molecules, such as N-Cadherin and NCAM (Neural Cell Adhesion Molecule), and NMDA (N-Methyl-D-Aspartate)-type glutamate receptors. Thus, it has been hypothesized that some drugs available for manipulating the central nervous system(CNS) may also act on the pancreatic ß- cells and may be of use for T2DM and MODY treatment. NMDA receptors represent key targets for drugs against several neuronal diseases with excitotoxicity as a contributing mechanism, such as Parkinson's and Alzheimer disease, as well as for the therapy of CNS-controlled disease symptoms, such as coughing.

Glutamate NMDA receptors are transmembrane, excitatory cell surface receptors at the level of the CNS and pancreatic islets. NMDA antagonists thus exert a preponderantly antiexcitatory effect on the CNS and decrease the central activation of the adrenal gland. This potentially leads to indirect effects on pancreatic cells and insulin secretion, but even direct effects on pancreatic ß-cells have been suggested by the antagonism of pancreatic NMDA receptors.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with a diagnosis of type 2 diabetes mellitus according to ADA criteria at least 4 months prior to screening
* Medical history without major pathology (with the exception of type 2 diabetes)
* On a stable regimen of metformin monotherapy for at least 3 months
* Body mass index (BMI) between 25 and 35kg/m2, both inclusive
* HbA1c ≥ 6.5 and <7.5%
* A male subject who is sexually active and not surgically sterilised, must agree to use adequate contraceptive methods from the time of first study drug administration until 90 days after last dosing.
* Ability and willingness to abstain from grapefruit juice (and all grapefruit containing products) throughout the study starting 24 hours prior to first study drug administration and from alcohol, methylxanthine-containing beverages or food (coffee, tea, Coke, chocolate, "power drinks"), tobacco products and from engaging in strenuous physical activity from 24 hours prior to each admission until discharge from the unit.

Exclusion Criteria:

* Subjects with type 1 diabetes, maturity onset diabetes of the young (MODY) or secondary forms of diabetes such as due to pancreatitis
* Current or previous treatment with insulin therapy (except for treatment within a clinical trial, for surgical procedures or during an acute illness for 7 days and more than 14 days before the first administration of study drug)
* Treatment with any hypoglycaemic medication other than metformin within the three months prior to screening
* Subjects with any severe medical or surgical history of conditions likely to confound study assessments or study endpoints, for example but not limited to haemoglobinopathies, inflammatory bowel disease, cystic fibrosis, bariatric surgery and/or any surgery shortening the intestine, history of galactose intolerance, lactose- or glucose-galactose-malabsorption
* Serious respiratory, serious and/or unstable coronary heart disease (unstable angina, myocardial infarction within the preceding 6 months), congestive heart failure of New York Heart Association Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnoea), second/third degree heart block, superior vena cava syndrome, uncontrolled hypertension, history of congenital QT-syndrome within family, history of stroke (within the preceding 6 months) or serious peripheral vascular disease
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (grade 3), left bundle branch block, or asymptomatic sustained ventricular tachycardia are not allowed
* Marked diabetic complications: severe autonomic or sensory neuropathy including gastroparesis; proliferative retinopathy
* Any respiratory disease leading to respiratory insufficiency and/or depression including but not limited to: asthma bronchiale, chronic obstructive pulmonary disease.
* Clinically significant vital signs including known bradycardia with pulse rate < 55/min or 12-lead ECG findings including pre-treatment QTc > 420 msec (if the ECG shows a QTc value of > 420 ms, two further ECGs will be repeated within the next 30 minutes, at least 2 minutes apart, with the mean value of these 3 consecutive ECGs being conclusive).
* History of or current prostata hyperplasia
* History of or current narrow angle glaucoma
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis or coagulation screening tests, as judged by the Investigator
* Moderate or severe renal dysfunction defined as a calculated GFR < 70 ml/min using the Cockcroft-Gault calculation
* Clinical or laboratory evidence of hepatic dysfunction or disease; laboratory evidence defined as any of the following parameters: alkaline phosphatase > 2x upper limit of normal (ULN), ALT > 2x ULN, AST > 2x ULN or bilirubin > 3x ULN. Isolated mild rise in bilirubin considered to be due to Gilbert's condition is allowed
* Uncontrolled high blood pressure (DBP > 95 mmHg and/or SBP > 160 mmHg), unless clearly documented to be white-coat hypertension
* History of any psychiatric condition that might impair the subject's ability to understand or to comply with the requirements of the study or to provide informed consent
* History of relevant drug and/or food allergies or a history of severe anaphylactic reaction
* Smoking more than 5 cigarettes/cigars/pipes daily and not willing to abstain from any consume of tobacco products 24 hours prior to each admission until discharge
* Currently active or history of alcohol abuse (defined as an intake of more than 24 units of alcohol per week; one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits) or drug addiction (including soft drugs like cannabis products)
* Positive alcohol test at screening Use of concomitant medication which would confound study conduct
* Monoamine oxidase (MAO) inhibitors or selective serotonin reuptake inhibitors (SSRI) (Fluoxetine, Paroxetine), any other antipsychotic and antidepressant medication or drugs with depressant effects on the central nervous system.
* Antiarrhythmic therapy class IA (e.g. Chinidin, Disopyramide, Procainamide) and class III (e.g. Sotalol)
* Antihistaminic therapy (e.g. Astemizole, Terfenadine)
* Use of macrolide antibiotics (e.g. Erythromycin, Clarythromycin) and gyrase inhibitors (e.g. Sparfloxacin) Use of antimycotic therapy (e.g. Bupidin, Halofantrine, Cotrimoxazole, Pentamidine, Cisapride, Bepridil)
* Use of weight-loss agents
* Medications which have the potential to inhibit CYP450 2D6: Amiodarone, Chinidin, Haloperidol, Paroxetine, Propafenone, Thioridazine, Cimetidine and Ritonavir.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose (BG) concentration-time profile | from 1-3 hours post-dose (i.e. from 0-2 hours after an OGTT)

SECONDARY OUTCOMES:
Area under the blood glucose concentration-time profile | 0-1 hour post-dose (i.e. before starting the OGTT)
Adverse events | 5 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Alin O Stirban, MD, Principal Investigator — Profil Institute for Metabolic Research
Locations (1):
- Profil Institute for Metabolic Research, Neuss, North Rhine-Westphalia, Germany